CLINICAL TRIAL: NCT07222696
Title: Pilot Randomized Trial of Health Coaching for People With Rheumatoid Arthritis to Improve Mental Well-Being
Brief Title: Healthier: Health Coaching for People With Rheumatoid Arthritis to Improve Mental Well-Being
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25-05028875
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA
Keywords: Rheumatoid Arthritis; Peer Coaching; Health Coaching; Community-based Intervention; Mental Health; Pain and mood management
MeSH Terms: conditions — Arthritis, Rheumatoid; Psychological Well-Being; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthier (Experimental): Participants will have 9 telephone-delivered sessions, over a 9-12-week period, delivered by a peer coach (another person with RA). Data will be collected at baseline, midway through the intervention (after Session 4 of the intervention), 3 weeks after completion of the intervention, 6, 12, and 24 months after completion of the intervention using validated instruments.
  Interventions: Behavioral: Peer Coach
- Healthy Horizons (Active Comparator): Participants from will have 9 telephone-delivered sessions over a 9-12-week period delivered by a coach (a person without RA but who has a different chronic condition like osteoarthritis or diabetes). Data will be collected at baseline, midway through the intervention (after Session 4 of the intervention), 3 weeks after completion of the intervention, 6, 12, and 24 months after completion of the intervention using validated instruments.
  Interventions: Behavioral: Healthy Horizons

INTERVENTIONS:
Behavioral: Peer Coach — The method that will be used in this trial will be peer coaching. Peer coaches are lay individuals who themselves have the targeted chronic condition, that for the purpose of this study is people with RA, allowing people to identify with their peers and increase confidence that they too can achieve favorable outcomes. They will use components of CBT, mindfulness, and exercise material that have been effective in improving mental and physical health in patients with RA. The Healthier intervention is distinct from these others because it focuses on a high-priority symptom experienced by people with RA: chronic pain. It mobilizes a behavior that impacts numerous dimensions beyond pain, including mobility, mood, cardiovascular health, and mortality.
  Arms: Healthier
Behavioral: Healthy Horizons — Participants in the active comparator arm will have telephone calls with a coach that does not have rheumatoid arthritis and who will deliver a nine-session intervention on general health topics that are widely available including topics on nutrition and cancer awareness. These coaches will not use CBT, mindfulness or make any references to exercise or physical activity.
  Arms: Healthy Horizons

SUMMARY:
The goal of this clinical trial is to learn if peer coaching works to reduce levels of anxiety and/or depression in adults diagnosed with Rheumatoid Arthritis (RA). The main questions it aims to answer are: Do people with RA who complete the intervention with a peer coach have lower levels of anxiety and/or depression at 6 months from baseline? Do people with RA who complete the intervention with a peer coach have lower levels of anxiety and/or depression at 6 months compared to those in the control arm?

Researchers will compare the peer coaching intervention to an active-control arm (where people without RA coach participants on general health and nutrition topics) to see if peer coaching works to reduce anxiety and/or depression.

Participants will meet with a coach every week for 9 weeks and complete several surveys before, during and after the intervention

ELIGIBILITY:
Inclusion Criteria:

* Male or Female older than 18 years of age.
* Have a diagnosis of Rheumatoid Arthritis by a rheumatologist and currently taking a Disease-Modifying Anti-rheumatic drug ( Conventional Disease-Modifying Anti-rheumatic drug and/or Biological Disease-Modifying Anti-rheumatic drug)
* Have high levels of depression defined as PHQ-8 scores between 10 to 20, OR high levels of anxiety based on GAD-7 scores > 10
* Speaks English or Spanish
* Have access to the internet, a computer, and/or a smartphone
* Resides or lives in any state of the US, including Puerto Rico
* Willing to work with a peer coach or a coach

Exclusion Criteria:

* Having a rheumatic disease other than RA (e.g., psoriatic arthritis, gout, lupus)
* Nursing home resident
* History of dementia or severe cognitive decline
* Are currently bedbound
* Severe depression defined as PHQ-8 scores of >20.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Mean Scores in PHQ-8 at 6 months post intervention | Baseline and 6 months after completing the intervention (35 weeks after baseline)
  Patient Health Questionnaire-8 has a range 0-24, where a higher score means more distress. The questions ask about how often participants have been affected by certain events.
Difference in Mean Scores in PHQ-8 Between the Experimental Arm and the Active Control Arm at 6 Months Post Intervention | Six months post intervention completion (Approximately 35 weeks after baseline)
  Patient Health Questionnaire-8 has a range 0-24, where a higher score means more distress. The questions ask about how often participants have been affected by certain events. We will determine differences in mean scores in PHQ-8 between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Change from Baseline in Mean Scores in GAD-7 at 6 months post intervention | Baseline and 6 months after completing the intervention (35 weeks after baseline)
  General Anxiety Disorder-7 has a range 0-21, where a score of 0-4 means minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety and 15-21 severe anxiety. The questions ask about how often participants have been affected by certain events.
Difference in Mean Scores in GAD-7 Between the Experimental Arm and the Active Control Arm at 6 Months Post Intervention | Six months post intervention completion (35 weeks after baseline)
  General Anxiety Disorder-7 has a range 0-21, where a score of 0-4 means minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety and 15-21 severe anxiety. The questions ask about how often participants have been affected by certain events. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms,

SECONDARY OUTCOMES:
Change from Baseline in Mean Scores in PROMIS Pain Interference Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference has a range of T-scores typically from 40 to 80, where a higher score means greater interference of pain with daily activities. The questions ask about how often pain has affected aspects of life such as social, cognitive, emotional, physical, and recreational functioning.
Change from Baseline in Mean Scores in PROMIS Pain Interference at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference has a range of T-scores typically from 40 to 80, where a higher score means greater interference of pain with daily activities. The questions ask about how often pain has affected aspects of life such as social, cognitive, emotional, physical, and recreational functioning.
Change from Baseline in Mean Scores in PROMIS Pain Interference at 6 Months Post-Intervention Completion | Baseline, 6 months post intervention completion (35 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference has a range of T-scores typically from 40 to 80, where a higher score means greater interference of pain with daily activities. The questions ask about how often pain has affected aspects of life such as social, cognitive, emotional, physical, and recreational functioning.
Change from Baseline in Mean Scores in PROMIS Pain Interference at 12 Months Post-Intervention Completion | Baseline, 12 months post-intervention completion (61 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference has a range of T-scores typically from 40 to 80, where a higher score means greater interference of pain with daily activities. The questions ask about how often pain has affected aspects of life such as social, cognitive, emotional, physical, and recreational functioning.
Change from Baseline in Mean Scores in PROMIS Pain Interference at 24 Months Post-Intervention Completion | Baseline, 24 months post-intervention completion (113 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference has a range of T-scores typically from 40 to 80, where a higher score means greater interference of pain with daily activities. The questions ask about how often pain has affected aspects of life such as social, cognitive, emotional, physical, and recreational functioning.
Difference in Mean Scores in PROMIS Pain Interference Between the Experimental Arm and the Active Control Arm Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference has a range of T-scores typically from 40 to 80, where a higher score means greater interference of pain with daily activities. The questions ask about how often pain has affected aspects of life such as social, cognitive, emotional, physical, and recreational functioning. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Pain Interference Between the Experimental Arm and the Active Control Arm at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention(12 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference has a range of T-scores typically from 40 to 80, where a higher score means greater interference of pain with daily activities. The questions ask about how often pain has affected aspects of life such as social, cognitive, emotional, physical, and recreational functioning. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Pain Interference Between the Experimental Arm and the Active Control Arm at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference has a range of T-scores typically from 40 to 80, where a higher score means greater interference of pain with daily activities. The questions ask about how often pain has affected aspects of life such as social, cognitive, emotional, physical, and recreational functioning. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Pain Interference Between the Experimental Arm and the Active Control Arm at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference has a range of T-scores typically from 40 to 80, where a higher score means greater interference of pain with daily activities. The questions ask about how often pain has affected aspects of life such as social, cognitive, emotional, physical, and recreational functioning. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Pain Interference Between the Experimental Arm and the Active Control Arm at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference has a range of T-scores typically from 40 to 80, where a higher score means greater interference of pain with daily activities. The questions ask about how often pain has affected aspects of life such as social, cognitive, emotional, physical, and recreational functioning. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Change from Baseline in Mean Scores in PROMIS Sleep Disturbance Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance has a range of T-scores typically from 40 to 80, where a higher score means greater interference of poor sleep with daily functioning and well-being. The questions ask about how often sleep problems have affected aspects of life such as alertness, mood, concentration, and energy..
Change from Baseline in Mean Scores in PROMIS Sleep Disturbance at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance has a range of T-scores typically from 40 to 80, where a higher score means greater interference of poor sleep with daily functioning and well-being. The questions ask about how often sleep problems have affected aspects of life such as alertness, mood, concentration, and energy..
Change from Baseline in Mean Scores in PROMIS Sleep Disturbance at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance has a range of T-scores typically from 40 to 80, where a higher score means greater interference of poor sleep with daily functioning and well-being. The questions ask about how often sleep problems have affected aspects of life such as alertness, mood, concentration, and energy..
Change from Baseline in Mean Scores in PROMIS Sleep Disturbance at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance has a range of T-scores typically from 40 to 80, where a higher score means greater interference of poor sleep with daily functioning and well-being. The questions ask about how often sleep problems have affected aspects of life such as alertness, mood, concentration, and energy..
Change from Baseline in Mean Scores in PROMIS Sleep Disturbance at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance has a range of T-scores typically from 40 to 80, where a higher score means greater interference of poor sleep with daily functioning and well-being. The questions ask about how often sleep problems have affected aspects of life such as alertness, mood, concentration, and energy..
Difference in Mean Scores in PROMIS Sleep Disturbance Between the Experimental Arm and the Active Control Arm Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance has a range of T-scores typically from 40 to 80, where a higher score means greater interference of poor sleep with daily functioning and well-being. The questions ask about how often sleep problems have affected aspects of life such as alertness, mood, concentration, and energy. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Sleep Disturbance Between the Experimental Arm and the Active Control Arm at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance has a range of T-scores typically from 40 to 80, where a higher score means greater interference of poor sleep with daily functioning and well-being. The questions ask about how often sleep problems have affected aspects of life such as alertness, mood, concentration, and energy. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Sleep Disturbance Between the Experimental Arm and the Active Control Arm at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance has a range of T-scores typically from 40 to 80, where a higher score means greater interference of poor sleep with daily functioning and well-being. The questions ask about how often sleep problems have affected aspects of life such as alertness, mood, concentration, and energy. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Sleep Disturbance Between the Experimental Arm and the Active Control Arm at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion(61 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance has a range of T-scores typically from 40 to 80, where a higher score means greater interference of poor sleep with daily functioning and well-being. The questions ask about how often sleep problems have affected aspects of life such as alertness, mood, concentration, and energy. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Sleep Disturbance Between the Experimental Arm and the Active Control Arm at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance has a range of T-scores typically from 40 to 80, where a higher score means greater interference of poor sleep with daily functioning and well-being. The questions ask about how often sleep problems have affected aspects of life such as alertness, mood, concentration, and energy. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Change from Baseline in Mean Scores in Short Form-12 Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Short Form-12 Health Survey (SF-12) has a range of 0 to 100, where higher scores indicate better health status. The questions ask about physical and mental health over the past four weeks, covering areas such as physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being.
Change from Baseline in Mean Scores in Short Form-12 at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention(12 weeks after baseline)
  Short Form-12 Health Survey (SF-12) has a range of 0 to 100, where higher scores indicate better health status. The questions ask about physical and mental health over the past four weeks, covering areas such as physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being.
Change from Baseline in Mean Scores in Short Form-12 at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  Short Form-12 Health Survey (SF-12) has a range of 0 to 100, where higher scores indicate better health status. The questions ask about physical and mental health over the past four weeks, covering areas such as physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being.
Change from Baseline in Mean Scores in Short Form-12 at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  Short Form-12 Health Survey (SF-12) has a range of 0 to 100, where higher scores indicate better health status. The questions ask about physical and mental health over the past four weeks, covering areas such as physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being.
Change from Baseline in Mean Scores in Short Form-12 at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion(113 weeks after baseline)
  Short Form-12 Health Survey (SF-12) has a range of 0 to 100, where higher scores indicate better health status. The questions ask about physical and mental health over the past four weeks, covering areas such as physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being.
Difference in Mean Scores in Short-Form 12 Between the Experimental Arm and the Active Control Arm Midway Through the Intervention | Baseline, Midway Through the intervention(4 weeks after baseline)
  Short Form-12 Health Survey (SF-12) has a range of 0 to 100, where higher scores indicate better health status. The questions ask about physical and mental health over the past four weeks, covering areas such as physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms.
Difference in Mean Scores in Short-Form 12 Between the Experimental Arm and the Active Control Arm at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention(12 weeks after baseline)
  Short Form-12 Health Survey (SF-12) has a range of 0 to 100, where higher scores indicate better health status. The questions ask about physical and mental health over the past four weeks, covering areas such as physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms.
Difference in Mean Scores in Short-Form 12 Between the Experimental Arm and the Active Control Arm at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion(35 weeks after baseline)
  Short Form-12 Health Survey (SF-12) has a range of 0 to 100, where higher scores indicate better health status. The questions ask about physical and mental health over the past four weeks, covering areas such as physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms.
Difference in Mean Scores in Short-Form 12 Between the Experimental Arm and the Active Control Arm at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion(61 weeks after baseline)
  Short Form-12 Health Survey (SF-12) has a range of 0 to 100, where higher scores indicate better health status. The questions ask about physical and mental health over the past four weeks, covering areas such as physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms.
Difference in Mean Scores in Short-Form 12 Between the Experimental Arm and the Active Control Arm at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion(113 weeks after baseline)
  Short Form-12 Health Survey (SF-12) has a range of 0 to 100, where higher scores indicate better health status. The questions ask about physical and mental health over the past four weeks, covering areas such as physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms.
Change from Baseline in Mean Scores in PROMIS Physical Function Midway Through the Intervention | Baseline, Midway Through the Intervention (4 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function has a range of T-scores typically from 20 to 80, where a higher score means better physical functioning. The questions ask about the ability to perform everyday activities such as walking, climbing stairs, carrying groceries, or engaging in recreational activities.
Change from Baseline in Mean Scores in PROMIS Physical Function at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention(12 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function has a range of T-scores typically from 20 to 80, where a higher score means better physical functioning. The questions ask about the ability to perform everyday activities such as walking, climbing stairs, carrying groceries, or engaging in recreational activities.
Change from Baseline in Mean Scores in PROMIS Physical Function at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function has a range of T-scores typically from 20 to 80, where a higher score means better physical functioning. The questions ask about the ability to perform everyday activities such as walking, climbing stairs, carrying groceries, or engaging in recreational activities.
Change from Baseline in Mean Scores in PROMIS Physical Function at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function has a range of T-scores typically from 20 to 80, where a higher score means better physical functioning. The questions ask about the ability to perform everyday activities such as walking, climbing stairs, carrying groceries, or engaging in recreational activities.
Change from Baseline in Mean Scores in PROMIS Physical Function at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function has a range of T-scores typically from 20 to 80, where a higher score means better physical functioning. The questions ask about the ability to perform everyday activities such as walking, climbing stairs, carrying groceries, or engaging in recreational activities.
Difference in Mean Scores in PROMIS Physical Function Between the Experimental Arm and the Active Control Arm Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function has a range of T-scores typically from 20 to 80, where a higher score means better physical functioning. The questions ask about the ability to perform everyday activities such as walking, climbing stairs, carrying groceries, or engaging in recreational activities. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Physical Function Between the Experimental Arm and the Active Control Arm at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention(12 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function has a range of T-scores typically from 20 to 80, where a higher score means better physical functioning. The questions ask about the ability to perform everyday activities such as walking, climbing stairs, carrying groceries, or engaging in recreational activities. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Physical Function Between the Experimental Arm and the Active Control Arm at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function has a range of T-scores typically from 20 to 80, where a higher score means better physical functioning. The questions ask about the ability to perform everyday activities such as walking, climbing stairs, carrying groceries, or engaging in recreational activities. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Physical Function Between the Experimental Arm and the Active Control Arm at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function has a range of T-scores typically from 20 to 80, where a higher score means better physical functioning. The questions ask about the ability to perform everyday activities such as walking, climbing stairs, carrying groceries, or engaging in recreational activities. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PROMIS Physical Function Between the Experimental Arm and the Active Control Arm at 24 Months Post-Intervention Completionn | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function has a range of T-scores typically from 20 to 80, where a higher score means better physical functioning. The questions ask about the ability to perform everyday activities such as walking, climbing stairs, carrying groceries, or engaging in recreational activities. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Change from Baseline in Mean Scores in Lubben Social Isolation Midway Through the Intervention | Baseline, Midway through the intervention( 4 weeks after baseline)
  Lubben Social Isolation or Lubben Social Network Scale (LSNS-6) has a range of 0 to 30, where higher scores indicate stronger social connectedness and lower risk of isolation. The questions ask about the number of relatives and friends with whom participants have regular contact, feel close to, or can call on for help.
Change from Baseline in Mean Scores in Lubben Social Isolation at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention( 12 weeks after baseline)
  Lubben Social Isolation or Lubben Social Network Scale (LSNS-6) has a range of 0 to 30, where higher scores indicate stronger social connectedness and lower risk of isolation. The questions ask about the number of relatives and friends with whom participants have regular contact, feel close to, or can call on for help.
Change from Baseline in Mean Scores in Lubben Social Isolation at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion( 35 weeks after baseline)
  Lubben Social Isolation or Lubben Social Network Scale (LSNS-6) has a range of 0 to 30, where higher scores indicate stronger social connectedness and lower risk of isolation. The questions ask about the number of relatives and friends with whom participants have regular contact, feel close to, or can call on for help.
Change from Baseline in Mean Scores in Lubben Social Isolation at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion( 61 weeks after baseline)
  Lubben Social Isolation or Lubben Social Network Scale (LSNS-6) has a range of 0 to 30, where higher scores indicate stronger social connectedness and lower risk of isolation. The questions ask about the number of relatives and friends with whom participants have regular contact, feel close to, or can call on for help.
Change from Baseline in Mean Scores in Lubben Social Isolation at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion( 113 weeks after baseline)
  Lubben Social Isolation or Lubben Social Network Scale (LSNS-6) has a range of 0 to 30, where higher scores indicate stronger social connectedness and lower risk of isolation. The questions ask about the number of relatives and friends with whom participants have regular contact, feel close to, or can call on for help.
Difference in Mean Scores in Lubben Social Isolation Between the Experimental Arm and the Active Control Arm Midway Through the Intervention | Baseline, Midway through the intervention(4 weeks after baseline)
  Lubben Social Isolation or Lubben Social Network Scale (LSNS-6) has a range of 0 to 30, where higher scores indicate stronger social connectedness and lower risk of isolation. The questions ask about the number of relatives and friends with whom participants have regular contact, feel close to, or can call on for help. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Lubben Social Isolation Between the Experimental Arm and the Active Control Arm at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention(12 weeks after baseline)
  Lubben Social Isolation or Lubben Social Network Scale (LSNS-6) has a range of 0 to 30, where higher scores indicate stronger social connectedness and lower risk of isolation. The questions ask about the number of relatives and friends with whom participants have regular contact, feel close to, or can call on for help. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Lubben Social Isolation Between the Experimental Arm and the Active Control Arm at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion(35 weeks after baseline)
  Lubben Social Isolation or Lubben Social Network Scale (LSNS-6) has a range of 0 to 30, where higher scores indicate stronger social connectedness and lower risk of isolation. The questions ask about the number of relatives and friends with whom participants have regular contact, feel close to, or can call on for help. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Lubben Social Isolation Between the Experimental Arm and the Active Control Arm at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion(61 weeks after baseline)
  Lubben Social Isolation or Lubben Social Network Scale (LSNS-6) has a range of 0 to 30, where higher scores indicate stronger social connectedness and lower risk of isolation. The questions ask about the number of relatives and friends with whom participants have regular contact, feel close to, or can call on for help. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Lubben Social Isolation Between the Experimental Arm and the Active Control Arm 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion(113 weeks after baseline)
  Lubben Social Isolation or Lubben Social Network Scale (LSNS-6) has a range of 0 to 30, where higher scores indicate stronger social connectedness and lower risk of isolation. The questions ask about the number of relatives and friends with whom participants have regular contact, feel close to, or can call on for help. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Change from Baseline in Mean Scores in Cohen Stress Scale Midway Through the Intervention | Baseline, Midway through the intervention(4 weeks after baseline)
  Cohen's Perceived Stress Scale (PSS) has a range of 0 to 40, where higher scores indicate greater perceived stress. The questions ask about how often participants have felt stressed, overwhelmed, or unable to control important aspects of their life over the past month. Scores of 0-13 are considered low stress, 14-26 moderate stress, and 27-40 high stress
Change from Baseline in Mean Scores in Cohen Stress Scale at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention(12 weeks after baseline)
  Cohen's Perceived Stress Scale (PSS) has a range of 0 to 40, where higher scores indicate greater perceived stress. The questions ask about how often participants have felt stressed, overwhelmed, or unable to control important aspects of their life over the past month. Scores of 0-13 are considered low stress, 14-26 moderate stress, and 27-40 high stress
Change from Baseline in Mean Scores in Cohen Stress Scale at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion(35 weeks after baseline)
  Cohen's Perceived Stress Scale (PSS) has a range of 0 to 40, where higher scores indicate greater perceived stress. The questions ask about how often participants have felt stressed, overwhelmed, or unable to control important aspects of their life over the past month. Scores of 0-13 are considered low stress, 14-26 moderate stress, and 27-40 high stress
Change from Baseline in Mean Scores in Cohen Stress Scale at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion(61 weeks after baseline)
  Cohen's Perceived Stress Scale (PSS) has a range of 0 to 40, where higher scores indicate greater perceived stress. The questions ask about how often participants have felt stressed, overwhelmed, or unable to control important aspects of their life over the past month. Scores of 0-13 are considered low stress, 14-26 moderate stress, and 27-40 high stress
Change from Baseline in Mean Scores in Cohen Stress Scale at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion(113 weeks after baseline)
  Cohen's Perceived Stress Scale (PSS) has a range of 0 to 40, where higher scores indicate greater perceived stress. The questions ask about how often participants have felt stressed, overwhelmed, or unable to control important aspects of their life over the past month. Scores of 0-13 are considered low stress, 14-26 moderate stress, and 27-40 high stress
Difference in Mean Scores in Cohen Stress Scale Between the Experimental Arm and the Active Control Arm Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Cohen's Perceived Stress Scale (PSS) has a range of 0 to 40, where higher scores indicate greater perceived stress. The questions ask about how often participants have felt stressed, overwhelmed, or unable to control important aspects of their life over the past month. Scores of 0-13 are considered low stress, 14-26 moderate stress, and 27-40 high stress. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Cohen Stress Scale Between the Experimental Arm and the Active Control Arm at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  Cohen's Perceived Stress Scale (PSS) has a range of 0 to 40, where higher scores indicate greater perceived stress. The questions ask about how often participants have felt stressed, overwhelmed, or unable to control important aspects of their life over the past month. Scores of 0-13 are considered low stress, 14-26 moderate stress, and 27-40 high stress. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Cohen Stress Scale Between the Experimental Arm and the Active Control Arm at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  Cohen's Perceived Stress Scale (PSS) has a range of 0 to 40, where higher scores indicate greater perceived stress. The questions ask about how often participants have felt stressed, overwhelmed, or unable to control important aspects of their life over the past month. Scores of 0-13 are considered low stress, 14-26 moderate stress, and 27-40 high stress. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Cohen Stress Scale Between the Experimental Arm and the Active Control Arm at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  Cohen's Perceived Stress Scale (PSS) has a range of 0 to 40, where higher scores indicate greater perceived stress. The questions ask about how often participants have felt stressed, overwhelmed, or unable to control important aspects of their life over the past month. Scores of 0-13 are considered low stress, 14-26 moderate stress, and 27-40 high stress. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Cohen Stress Scale Between the Experimental Arm and the Active Control Arm at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  Cohen's Perceived Stress Scale (PSS) has a range of 0 to 40, where higher scores indicate greater perceived stress. The questions ask about how often participants have felt stressed, overwhelmed, or unable to control important aspects of their life over the past month. Scores of 0-13 are considered low stress, 14-26 moderate stress, and 27-40 high stress. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Change from Baseline in Mean Scores in UCLA Loneliness Scale Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  UCLA Loneliness Scale has a range of 20 to 80, where higher scores indicate greater loneliness. The questions ask about how often participants feel lacking in companionship, left out, or isolated from others.
Change from Baseline in Mean Scores in UCLA Loneliness Scale at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  UCLA Loneliness Scale has a range of 20 to 80, where higher scores indicate greater loneliness. The questions ask about how often participants feel lacking in companionship, left out, or isolated from others.
Change from Baseline in Mean Scores in UCLA Loneliness Scale at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  UCLA Loneliness Scale has a range of 20 to 80, where higher scores indicate greater loneliness. The questions ask about how often participants feel lacking in companionship, left out, or isolated from others.
Change from Baseline in Mean Scores in UCLA Loneliness Scale at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  UCLA Loneliness Scale has a range of 20 to 80, where higher scores indicate greater loneliness. The questions ask about how often participants feel lacking in companionship, left out, or isolated from others.
Change from Baseline in Mean Scores in UCLA Loneliness Scale at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  UCLA Loneliness Scale has a range of 20 to 80, where higher scores indicate greater loneliness. The questions ask about how often participants feel lacking in companionship, left out, or isolated from others.
Difference in Mean Scores in UCLA Loneliness Scale Between the Experimental Arm and the Active Control Arm Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  UCLA Loneliness Scale has a range of 20 to 80, where higher scores indicate greater loneliness. The questions ask about how often participants feel lacking in companionship, left out, or isolated from others. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in UCLA Loneliness Scale Between the Experimental Arm and the Active Control Arm at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  UCLA Loneliness Scale has a range of 20 to 80, where higher scores indicate greater loneliness. The questions ask about how often participants feel lacking in companionship, left out, or isolated from others. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in UCLA Loneliness Scale Between the Experimental Arm and the Active Control Arm at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  UCLA Loneliness Scale has a range of 20 to 80, where higher scores indicate greater loneliness. The questions ask about how often participants feel lacking in companionship, left out, or isolated from others. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in UCLA Loneliness Scale Between the Experimental Arm and the Active Control Arm at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  UCLA Loneliness Scale has a range of 20 to 80, where higher scores indicate greater loneliness. The questions ask about how often participants feel lacking in companionship, left out, or isolated from others. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in UCLA Loneliness Scale Between the Experimental Arm and the Active Control Arm at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  UCLA Loneliness Scale has a range of 20 to 80, where higher scores indicate greater loneliness. The questions ask about how often participants feel lacking in companionship, left out, or isolated from others. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Change from Baseline in Mean Scores in Pain Self-Efficacy Questionnaire Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Pain Self-Efficacy Questionnaire (PSEQ) has a range of 0 to 60, where higher scores indicate greater confidence in the ability to perform activities despite pain. The questions ask about how certain participants feel they can manage daily tasks, work, and social activities while living with pain.
Change from Baseline in Mean Scores in Pain Self-Efficacy Questionnaire at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  Pain Self-Efficacy Questionnaire (PSEQ) has a range of 0 to 60, where higher scores indicate greater confidence in the ability to perform activities despite pain. The questions ask about how certain participants feel they can manage daily tasks, work, and social activities while living with pain.
Change from Baseline in Mean Scores in Pain Self-Efficacy Questionnaire at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  Pain Self-Efficacy Questionnaire (PSEQ) has a range of 0 to 60, where higher scores indicate greater confidence in the ability to perform activities despite pain. The questions ask about how certain participants feel they can manage daily tasks, work, and social activities while living with pain.
Change from Baseline in Mean Scores in Pain Self-Efficacy Questionnaire at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  Pain Self-Efficacy Questionnaire (PSEQ) has a range of 0 to 60, where higher scores indicate greater confidence in the ability to perform activities despite pain. The questions ask about how certain participants feel they can manage daily tasks, work, and social activities while living with pain.
Change from Baseline in Mean Scores in Pain Self-Efficacy Questionnaire at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  Pain Self-Efficacy Questionnaire (PSEQ) has a range of 0 to 60, where higher scores indicate greater confidence in the ability to perform activities despite pain. The questions ask about how certain participants feel they can manage daily tasks, work, and social activities while living with pain.
Difference in Mean Scores in Pain Self-Efficacy Questionnaire Between the Experimental Arm and the Active Control Arm Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Pain Self-Efficacy Questionnaire (PSEQ) has a range of 0 to 60, where higher scores indicate greater confidence in the ability to perform activities despite pain. The questions ask about how certain participants feel they can manage daily tasks, work, and social activities while living with pain. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Pain Self-Efficacy Questionnaire Between the Experimental Arm and the Active Control Arm at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  Pain Self-Efficacy Questionnaire (PSEQ) has a range of 0 to 60, where higher scores indicate greater confidence in the ability to perform activities despite pain. The questions ask about how certain participants feel they can manage daily tasks, work, and social activities while living with pain. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Pain Self-Efficacy Questionnaire Between the Experimental Arm and the Active Control Arm at 6 Months Post-Intervention Completion | Baseline, 6 Months Post-Intervention Completion (35 weeks after baseline)
  Pain Self-Efficacy Questionnaire (PSEQ) has a range of 0 to 60, where higher scores indicate greater confidence in the ability to perform activities despite pain. The questions ask about how certain participants feel they can manage daily tasks, work, and social activities while living with pain. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Pain Self-Efficacy Questionnaire Between the Experimental Arm and the Active Control Arm at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  Pain Self-Efficacy Questionnaire (PSEQ) has a range of 0 to 60, where higher scores indicate greater confidence in the ability to perform activities despite pain. The questions ask about how certain participants feel they can manage daily tasks, work, and social activities while living with pain. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in Pain Self-Efficacy Questionnaire Between the Experimental Arm and the Active Control Arm at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  Pain Self-Efficacy Questionnaire (PSEQ) has a range of 0 to 60, where higher scores indicate greater confidence in the ability to perform activities despite pain. The questions ask about how certain participants feel they can manage daily tasks, work, and social activities while living with pain. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Change from Baseline in Mean Scores in PHQ-8 Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Patient Health Questionnaire-8 has a range 0-24, where a higher score means more distress. The questions ask about how often participants have been affected by certain events.
Change from Baseline in Mean Scores in PHQ-8 at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  Patient Health Questionnaire-8 has a range 0-24, where a higher score means more distress. The questions ask about how often participants have been affected by certain events.
Change from Baseline in Mean Scores in PHQ-8 at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  Patient Health Questionnaire-8 has a range 0-24, where a higher score means more distress. The questions ask about how often participants have been affected by certain events.
Change from Baseline in Mean Scores in PHQ-8 at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  Patient Health Questionnaire-8 has a range 0-24, where a higher score means more distress. The questions ask about how often participants have been affected by certain events.
Difference in Mean Scores in PHQ-8 Between the Experimental Arm and the Active Control Arm Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  Patient Health Questionnaire-8 has a range 0-24, where a higher score means more distress. The questions ask about how often participants have been affected by certain events. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PHQ-8 Between the Experimental Arm and the Active Control Arm at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  Patient Health Questionnaire-8 has a range 0-24, where a higher score means more distress. The questions ask about how often participants have been affected by certain events. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PHQ-8 Between the Experimental Arm and the Active Control Arm at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  Patient Health Questionnaire-8 has a range 0-24, where a higher score means more distress. The questions ask about how often participants have been affected by certain events. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in PHQ-8 Between the Experimental Arm and the Active Control Arm at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  Patient Health Questionnaire-8 has a range 0-24, where a higher score means more distress. The questions ask about how often participants have been affected by certain events. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Change from Baseline in Mean Scores in GAD-7 Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  General Anxiety Disorder-7 has a range 0-21, where a score of 0-4 means minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety and 15-21 severe anxiety. The questions ask about how often participants have been affected by certain events.
Change from Baseline in Mean Scores in GAD-7 at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  General Anxiety Disorder-7 has a range 0-21, where a score of 0-4 means minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety and 15-21 severe anxiety. The questions ask about how often participants have been affected by certain events.
Change from Baseline in Mean Scores in GAD-7 at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  General Anxiety Disorder-7 has a range 0-21, where a score of 0-4 means minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety and 15-21 severe anxiety. The questions ask about how often participants have been affected by certain events.
Change from Baseline in Mean Scores in GAD-7 at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion(113 weeks after baseline)
  General Anxiety Disorder-7 has a range 0-21, where a score of 0-4 means minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety and 15-21 severe anxiety. The questions ask about how often participants have been affected by certain events.
Difference in Mean Scores in GAD-7 Between the Experimental Arm and the Active Control Arm Midway Through the Intervention | Baseline, Midway through the intervention (4 weeks after baseline)
  General Anxiety Disorder-7 has a range 0-21, where a score of 0-4 means minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety and 15-21 severe anxiety. The questions ask about how often participants have been affected by certain events. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in GAD-7 Between the Experimental Arm and the Active Control Arm at 3 Weeks Post-Intervention | Baseline, 3 Weeks Post-Intervention (12 weeks after baseline)
  General Anxiety Disorder-7 has a range 0-21, where a score of 0-4 means minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety and 15-21 severe anxiety. The questions ask about how often participants have been affected by certain events. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in GAD-7 Between the Experimental Arm and the Active Control Arm at 12 Months Post-Intervention Completion | Baseline, 12 Months Post-Intervention Completion (61 weeks after baseline)
  General Anxiety Disorder-7 has a range 0-21, where a score of 0-4 means minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety and 15-21 severe anxiety. The questions ask about how often participants have been affected by certain events. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms
Difference in Mean Scores in GAD-7 Between the Experimental Arm and the Active Control Arm at 24 Months Post-Intervention Completion | Baseline, 24 Months Post-Intervention Completion (113 weeks after baseline)
  General Anxiety Disorder-7 has a range 0-21, where a score of 0-4 means minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety and 15-21 severe anxiety. The questions ask about how often participants have been affected by certain events. We will determine differences in mean scores between the experimental arm and the active control arm to establish whether or not there is a clinical significant difference between arms

CONTACTS AND LOCATIONS:
Overall Officials: Iris Y Navarro-Millán, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared upon reasonable request and with a proposal.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 9 months following the last data collection and ending 72 months following publication.
Access Criteria: Investigators may request data for meta-analysis. Proposals should be directed to yin9003@med.cornell.edu to gain access, data requestors will need to sign a data access agreement upon data availability.

REFERENCES:
- [Background] Little RJ, Wang Y. Pattern-mixture models for multivariate incomplete data with covariates. Biometrics. 1996 Mar;52(1):98-111. PMID 8934587
- [Background] Royston P, White IR. Multiple imputation by chained equations (MICE): implementation in Stata. Journal of statistical software. 2011;45:1-20
- [Background] McCurry SM, Von Korff M, Vitiello MV, Saunders K, Balderson BH, Moore AL, Rybarczyk BD. Frequency of comorbid insomnia, pain, and depression in older adults with osteoarthritis: predictors of enrollment in a randomized treatment trial. J Psychosom Res. 2011 Nov;71(5):296-9. doi: 10.1016/j.jpsychores.2011.05.012. Epub 2011 Jul 1. PMID 21999972
- [Background] Vasiliadis HM, Chudzinski V, Gontijo-Guerra S, Preville M. Screening instruments for a population of older adults: The 10-item Kessler Psychological Distress Scale (K10) and the 7-item Generalized Anxiety Disorder Scale (GAD-7). Psychiatry Res. 2015 Jul 30;228(1):89-94. doi: 10.1016/j.psychres.2015.04.019. Epub 2015 Apr 23. PMID 25956759
- [Background] Osman A, Barrios FX, Kopper BA, Hauptmann W, Jones J, O'Neill E. Factor structure, reliability, and validity of the Pain Catastrophizing Scale. J Behav Med. 1997 Dec;20(6):589-605. doi: 10.1023/a:1025570508954. PMID 9429990
- [Background] Toussaint A, Husing P, Gumz A, Wingenfeld K, Harter M, Schramm E, Lowe B. Sensitivity to change and minimal clinically important difference of the 7-item Generalized Anxiety Disorder Questionnaire (GAD-7). J Affect Disord. 2020 Mar 15;265:395-401. doi: 10.1016/j.jad.2020.01.032. Epub 2020 Jan 15. PMID 32090765
- [Background] Kounali D, Button KS, Lewis G, Gilbody S, Kessler D, Araya R, Duffy L, Lanham P, Peters TJ, Wiles N, Lewis G. How much change is enough? Evidence from a longitudinal study on depression in UK primary care. Psychol Med. 2022 Jul;52(10):1875-1882. doi: 10.1017/S0033291720003700. Epub 2020 Nov 3. PMID 33138872
- [Background] Bauer-Staeb C, Kounali DZ, Welton NJ, Griffith E, Wiles NJ, Lewis G, Faraway JJ, Button KS. Effective dose 50 method as the minimal clinically important difference: Evidence from depression trials. J Clin Epidemiol. 2021 Sep;137:200-208. doi: 10.1016/j.jclinepi.2021.04.002. Epub 2021 Apr 20. PMID 33892086
- [Background] Safford MM, Cummings DM, Halladay JR, Shikany JM, Richman J, Oparil S, Hollenberg J, Adams A, Anabtawi M, Andreae L, Baquero E, Bryan J, Sanders-Clark D, Johnson E, Richman E, Soroka O, Tillman J, Cherrington AL. Practice Facilitation and Peer Coaching for Uncontrolled Hypertension Among Black Individuals: A Randomized Clinical Trial. JAMA Intern Med. 2024 May 1;184(5):538-546. doi: 10.1001/jamainternmed.2024.0047. PMID 38497987
- [Background] Safford MM, Andreae S, Cherrington AL, Martin MY, Halanych J, Lewis M, Patel A, Johnson E, Clark D, Gamboa C, Richman JS. Peer Coaches to Improve Diabetes Outcomes in Rural Alabama: A Cluster Randomized Trial. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S18-26. doi: 10.1370/afm.1798. PMID 26304967
- [Background] Richman JS, Andreae S, Safford MM. Challenges of Prolonged Follow-up and Temporal Imbalance in Pragmatic Trials: Analysis of the ENCOURAGE Trial. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S66-72. doi: 10.1370/afm.1790. PMID 26304974
- [Background] Guideline Development Panel for the Treatment of Depressive Disorders. Summary of the clinical practice guideline for the treatment of depression across three age cohorts. Am Psychol. 2022 Sep;77(6):770-780. doi: 10.1037/amp0000904. Epub 2021 Nov 29. PMID 34843274
- [Background] Salvi J. Calculated Decisions: Columbia-Suicide Severity Rating Scale (C-SSRS). Emerg Med Pract. 2019 May 1;21(5):CD3-4. PMID 31039299
- [Background] Pedersen JK, Wang L, Risbo N, Pedersen AB, Andersen K, Ellingsen T. Mortality in patients with incident rheumatoid arthritis and depression: a Danish cohort study of 11 071 patients and 55 355 comparators. Rheumatology (Oxford). 2024 Mar 1;63(3):680-688. doi: 10.1093/rheumatology/kead259. PMID 37252810
- [Background] Heidari P, Cross W, Crawford K. Do out-of-pocket costs affect medication adherence in adults with rheumatoid arthritis? A systematic review. Semin Arthritis Rheum. 2018 Aug;48(1):12-21. doi: 10.1016/j.semarthrit.2017.12.010. Epub 2018 Jan 8. PMID 29496225
- [Background] Barton JL, Trupin L, Schillinger D, Gansky SA, Tonner C, Margaretten M, Chernitskiy V, Graf J, Imboden J, Yelin E. Racial and ethnic disparities in disease activity and function among persons with rheumatoid arthritis from university-affiliated clinics. Arthritis Care Res (Hoboken). 2011 Sep;63(9):1238-46. doi: 10.1002/acr.20525. PMID 21671414
- [Background] Martin A, Chilton J, Paasche C, Nabatkhorian N, Gortler H, Cohenmehr E, Weller I, Amsalem D, Neary S. Shared Living Experiences by Physicians have a Positive Impact on Mental Health Attitudes and Stigma among Medical Students: A Mixed-Methods Study. J Med Educ Curric Dev. 2020 Oct 26;7:2382120520968072. doi: 10.1177/2382120520968072. eCollection 2020 Jan-Dec. PMID 33195803
- [Background] Moskalenko MY, Hadjistavropoulos HD, Katapally TR. Barriers to patient interest in internet-based cognitive behavioral therapy: Informing e-health policies through quantitative analysis. Health Policy and Technology. 2020/06/01/ 2020;9(2):139-145. https://doi.org/10.1016/j.hlpt.2020.04.004
- [Background] Wells MJ, Owen JJ, McCray LW, Bishop LB, Eells TD, Brown GK, Richards D, Thase ME, Wright JH. Computer-Assisted Cognitive-Behavior Therapy for Depression in Primary Care: Systematic Review and Meta-Analysis. Prim Care Companion CNS Disord. 2018 Mar 1;20(2):17r02196. doi: 10.4088/PCC.17r02196. PMID 29570963
- [Background] Rost T, Stein J, Lobner M, Kersting A, Luck-Sikorski C, Riedel-Heller SG. User Acceptance of Computerized Cognitive Behavioral Therapy for Depression: Systematic Review. J Med Internet Res. 2017 Sep 13;19(9):e309. doi: 10.2196/jmir.7662. PMID 28903893
- [Background] Carlbring P, Andersson G, Cuijpers P, Riper H, Hedman-Lagerlof E. Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: an updated systematic review and meta-analysis. Cogn Behav Ther. 2018 Jan;47(1):1-18. doi: 10.1080/16506073.2017.1401115. Epub 2017 Dec 7. PMID 29215315
- [Background] Proudfoot J, Ryden C, Everitt B, Shapiro DA, Goldberg D, Mann A, Tylee A, Marks I, Gray JA. Clinical efficacy of computerised cognitive-behavioural therapy for anxiety and depression in primary care: randomised controlled trial. Br J Psychiatry. 2004 Jul;185:46-54. doi: 10.1192/bjp.185.1.46. PMID 15231555
- [Background] Merry SN, Stasiak K, Shepherd M, Frampton C, Fleming T, Lucassen MF. The effectiveness of SPARX, a computerised self help intervention for adolescents seeking help for depression: randomised controlled non-inferiority trial. BMJ. 2012 Apr 18;344:e2598. doi: 10.1136/bmj.e2598. PMID 22517917
- [Background] Christensen H, Griffiths KM, Korten A. Web-based cognitive behavior therapy: analysis of site usage and changes in depression and anxiety scores. J Med Internet Res. 2002 Jan-Mar;4(1):e3. doi: 10.2196/jmir.4.1.e3. PMID 11956035
- [Background] Almohammed OA, Alsalem AA, Almangour AA, Alotaibi LH, Al Yami MS, Lai L. Antidepressants and health-related quality of life (HRQoL) for patients with depression: Analysis of the medical expenditure panel survey from the United States. PLoS One. 2022 Apr 20;17(4):e0265928. doi: 10.1371/journal.pone.0265928. eCollection 2022. PMID 35442954
- [Background] Young SD, Zhao M, Teiu K, Kwok J, Gill H, Gill N. A social-media based HIV prevention intervention using peer leaders. J Consum Health Internet. 2013 Oct 1;17(4):353-361. doi: 10.1080/15398285.2013.833445. PMID 24526928
- [Background] Fisher EB Jr, Strunk RC, Sussman LK, Arfken C, Sykes RK, Munro JM, Haywood S, Harrison D, Bascom S. Acceptability and feasibility of a community approach to asthma management: the Neighborhood Asthma Coalition (NAC). J Asthma. 1996;33(6):367-83. doi: 10.3109/02770909609068182. PMID 8968292
- [Background] Shah S, Peat JK, Mazurski EJ, Wang H, Sindhusake D, Bruce C, Henry RL, Gibson PG. Effect of peer led programme for asthma education in adolescents: cluster randomised controlled trial. BMJ. 2001 Mar 10;322(7286):583-5. doi: 10.1136/bmj.322.7286.583. PMID 11238152
- [Background] Horvath KJ, Oakes JM, Rosser BR, Danilenko G, Vezina H, Amico KR, Williams ML, Simoni J. Feasibility, acceptability and preliminary efficacy of an online peer-to-peer social support ART adherence intervention. AIDS Behav. 2013 Jul;17(6):2031-44. doi: 10.1007/s10461-013-0469-1. PMID 23553347
- [Background] Thom DH, Ghorob A, Hessler D, De Vore D, Chen E, Bodenheimer TA. Impact of peer health coaching on glycemic control in low-income patients with diabetes: a randomized controlled trial. Ann Fam Med. 2013 Mar-Apr;11(2):137-44. doi: 10.1370/afm.1443. PMID 23508600
- [Background] Tang TS, Funnell MM, Gillard M, Nwankwo R, Heisler M. The development of a pilot training program for peer leaders in diabetes: process and content. Diabetes Educ. 2011 Jan-Feb;37(1):67-77. doi: 10.1177/0145721710387308. Epub 2011 Jan 10. PMID 21220362
- [Background] Tang TS, Funnell MM, Gillard M, Nwankwo R, Heisler M. Training peers to provide ongoing diabetes self-management support (DSMS): results from a pilot study. Patient Educ Couns. 2011 Nov;85(2):160-8. doi: 10.1016/j.pec.2010.12.013. Epub 2011 Feb 2. PMID 21292425
- [Background] Tang TS, Funnell M, Sinco B, Piatt G, Palmisano G, Spencer MS, Kieffer EC, Heisler M. Comparative effectiveness of peer leaders and community health workers in diabetes self-management support: results of a randomized controlled trial. Diabetes Care. 2014 Jun;37(6):1525-34. doi: 10.2337/dc13-2161. Epub 2014 Apr 10. PMID 24722495
- [Background] Bandura A. Social cognitive theory: an agentic perspective. Annu Rev Psychol. 2001;52:1-26. doi: 10.1146/annurev.psych.52.1.1. PMID 11148297
- [Background] Shen B, Li Y, Du X, Chen H, Xu Y, Li H, Xu GY. Effects of cognitive behavioral therapy for patients with rheumatoid arthritis: a systematic review and meta-analysis. Psychol Health Med. 2020 Dec;25(10):1179-1191. doi: 10.1080/13548506.2020.1736312. Epub 2020 Mar 4. PMID 32129673
- [Background] Zhou B, Wang G, Hong Y, Xu S, Wang J, Yu H, Liu Y, Yu L. Mindfulness interventions for rheumatoid arthritis: A systematic review and meta-analysis. Complement Ther Clin Pract. 2020 May;39:101088. doi: 10.1016/j.ctcp.2020.101088. Epub 2020 Jan 11. PMID 31957665
- [Background] Andreae SJ, Andreae LJ, Richman JS, Cherrington AL, Safford MM. Peer-Delivered Cognitive Behavioral Training to Improve Functioning in Patients With Diabetes: A Cluster-Randomized Trial. Ann Fam Med. 2020 Jan;18(1):15-23. doi: 10.1370/afm.2469. PMID 31937528
- [Background] Benatti FB, Pedersen BK. Exercise as an anti-inflammatory therapy for rheumatic diseases-myokine regulation. Nat Rev Rheumatol. 2015 Feb;11(2):86-97. doi: 10.1038/nrrheum.2014.193. Epub 2014 Nov 25. PMID 25422002
- [Background] Rahman A, Malik A, Sikander S, Roberts C, Creed F. Cognitive behaviour therapy-based intervention by community health workers for mothers with depression and their infants in rural Pakistan: a cluster-randomised controlled trial. Lancet. 2008 Sep 13;372(9642):902-9. doi: 10.1016/S0140-6736(08)61400-2. PMID 18790313
- [Background] Meerwijk EL, Ford JM, Weiss SJ. Brain regions associated with psychological pain: implications for a neural network and its relationship to physical pain. Brain Imaging Behav. 2013 Mar;7(1):1-14. doi: 10.1007/s11682-012-9179-y. PMID 22660945
- [Background] Sheng J, Liu S, Wang Y, Cui R, Zhang X. The Link between Depression and Chronic Pain: Neural Mechanisms in the Brain. Neural Plast. 2017;2017:9724371. doi: 10.1155/2017/9724371. Epub 2017 Jun 19. PMID 28706741
- [Background] Bruce B, Fries JF, Murtagh KN. Health status disparities in ethnic minority patients with rheumatoid arthritis: a cross-sectional study. J Rheumatol. 2007 Jul;34(7):1475-9. Epub 2007 Jun 1. PMID 17552045
- [Background] Navarro-Millan I, Rajan M, Lui GE, Kern LM, Pinheiro LC, Safford MM, Sattui SE, Curtis JR. Racial and ethnic differences in medication use among beneficiaries of social security disability insurance with rheumatoid arthritis. Semin Arthritis Rheum. 2020 Oct;50(5):988-995. doi: 10.1016/j.semarthrit.2020.07.008. Epub 2020 Jul 23. PMID 32911290
- [Background] Yip K, Navarro-Millan I. Racial, ethnic, and healthcare disparities in rheumatoid arthritis. Curr Opin Rheumatol. 2021 Mar 1;33(2):117-121. doi: 10.1097/BOR.0000000000000782. PMID 33394602
- [Background] Alegria M, Chatterji P, Wells K, Cao Z, Chen CN, Takeuchi D, Jackson J, Meng XL. Disparity in depression treatment among racial and ethnic minority populations in the United States. Psychiatr Serv. 2008 Nov;59(11):1264-72. doi: 10.1176/ps.2008.59.11.1264. PMID 18971402
- [Background] Peterson S, Piercy J, Blackburn S, Sullivan E, Karyekar CS, Li N. The multifaceted impact of anxiety and depression on patients with rheumatoid arthritis. BMC Rheumatol. 2019 Oct 28;3:43. doi: 10.1186/s41927-019-0092-5. eCollection 2019. PMID 31673680
- [Background] Anyfanti P, Gavriilaki E, Pyrpasopoulou A, Triantafyllou G, Triantafyllou A, Chatzimichailidou S, Gkaliagkousi E, Aslanidis S, Douma S. Depression, anxiety, and quality of life in a large cohort of patients with rheumatic diseases: common, yet undertreated. Clin Rheumatol. 2016 Mar;35(3):733-9. doi: 10.1007/s10067-014-2677-0. Epub 2014 May 25. PMID 24859781
- [Background] Navarro-Millan I, Chen L, Greenberg JD, Pappas DA, Curtis JR. Predictors and persistence of new-onset clinical remission in rheumatoid arthritis patients. Semin Arthritis Rheum. 2013 Oct;43(2):137-43. doi: 10.1016/j.semarthrit.2013.02.002. Epub 2013 Jun 3. PMID 23742957
- [Background] Ni Mhuircheartaigh O, Crowson CS, Gabriel SE, Roger VL, Melton LJ 3rd, Amin S. Fragility Fractures Are Associated with an Increased Risk for Cardiovascular Events in Women and Men with Rheumatoid Arthritis: A Population-based Study. J Rheumatol. 2017 May;44(5):558-564. doi: 10.3899/jrheum.160651. Epub 2017 Jan 15. PMID 28089982